CLINICAL TRIAL: NCT02478333
Title: A Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of ALS-008176 in Healthy Japanese Adult Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of ALS-008176 in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR107180; 64041575RSV1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Healthy; ALS-008176; Japanese adult participants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALS-008176 (250 mg) or Placebo (Experimental): Participants will receive ALS-008176, 250 milligram (mg) or placebo oral suspension once on Day 1 under fasted conditions.
  Interventions: Drug: ALS-008176 (250 mg); Other: Placebo
- ALS-008176 (500 mg) or Placebo (Experimental): Participants will receive ALS-008176, 500 milligram (mg) or placebo oral suspension once on Day 1 under fasted conditions.
  Interventions: Drug: ALS-008176 (500 mg); Other: Placebo
- ALS-008176 (750 mg) or Placebo (Experimental): Participants will receive ALS-008176, 750 milligram (mg) or placebo oral suspension once on Day 1 under fasted conditions.
  Interventions: Drug: ALS-008176 (750 mg); Other: Placebo

INTERVENTIONS:
Drug: ALS-008176 (250 mg) — Participants will receive ALS-008176, 250 mg oral suspension once on Day 1 under fasted conditions.
  Arms: ALS-008176 (250 mg) or Placebo
Drug: ALS-008176 (500 mg) — Participants will receive ALS-008176, 500 mg oral suspension once on Day 1 under fasted conditions.
  Arms: ALS-008176 (500 mg) or Placebo
Drug: ALS-008176 (750 mg) — Participants will receive ALS-008176, 750 mg oral suspension once on Day 1 under fasted conditions.
  Arms: ALS-008176 (750 mg) or Placebo
Other: Placebo — Participants will receive placebo oral suspension once on Day 1 under fasted conditions.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ALS-008176 following oral administration of single ascending dose of ALS-008176 in healthy Japanese adult participants.

DETAILED DESCRIPTION:
This is a double-blind (test or experiment in which neither the person giving the treatment nor the patient knows which treatment the patient is receiving), placebo-controlled, randomized (study medication assigned to participants by chance) and single-center study of ALS-008176. The duration of study will be approximately 6 weeks for each participant. The study consists of 3 parts: Screening Phase (28 days before study commences on Day 1); double-blind Treatment Phase (single oral dose of ALS-008176 or placebo on Day 1 under fasted condition); and Follow up Phase (up to 14 days after study drug administration). All the eligible participants will be randomly assigned to receive either a single oral dose of ALS-008176 or placebo in each group. The planned doses will be escalated in a stepwise fashion if the safety and tolerability in the preceding dose is found acceptable. Participants in Group 1 will receive ALS-008176, 250 milligram (mg) or placebo, Group 2 will receive ALS-008176, 500 mg or placebo and Group 3 will receive ALS-008176, 750 mg or placebo. Study drug will be administered following a 10-hour overnight fast. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Pharmacokinetics of ALS-008176, ALS-008206, ALS-008112, and its metabolite ALS 008144 will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a Japanese participant whose parents and grandparents are Japanese as determined by the participant's verbal report
* Each participant must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A female participant must be either:

  1. Not of childbearing potential: postmenopausal [greater than (>) 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 International Units (IU)/ liter (L) (to be confirmed at Screening for all postmonopausal women)] OR
  2. Permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or otherwise incapable of becoming pregnant, OR c. If of childbearing potential and heterosexually active, practicing an effective method of birth control before entry and agree to continue to use two effective methods of contraception throughout the study and for at least 30 days after receiving the study drug
* Participant must be a non-smoker for at least one month prior to screening

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a past history of heart arrhythmias (extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Participant has creatinine clearance of lower than 70 millilitre (mL)/min
* Participant has taken any disallowed therapies as noted in protocol, Pre-study and Concomitant Therapy before the planned study drug
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The Cmax is the maximum observed plasma concentration of ALS 008176, ALS-008206, ALS-008112, and ALS-008144.
Time to Reach the Maximum Plasma Concentration (Tmax) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The Tmax is the time to reach the maximum observed plasma concentration of ALS 008176, ALS-008206, ALS-008112, and ALS-008144.
Time of Last Measurable Plasma Concentration (Tlast) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  Time of last measurable (non-below quantification limit [non-BQL]) plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The AUC (0-last) is the area under the plasma ALS 008176, ALS-008206, ALS-008112, and ALS-008144 concentration-time curve from time 0 to time of the last observed (non-BQL) quantifiable concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma ALS 008176, ALS-008206, ALS-008112, and ALS-008144 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed (non-BQL) quantifiable concentration and lambda(z) is elimination rate constant. Extrapolations of more than 20.00% of the total AUC are reported as approximations.
Percentage of Area Under the Plasma Concentration-Time Curve Obtained by Extrapolation (%AUC[infinity,ex]) | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The %AUC[infinity,ex] is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100, (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Apparent Initial Elimination Rate Constant (Lambda [alpha]) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The Lambda (alpha) determined by linear regression of the first elimination phase of the ln-linear plasma concentration-time curve.
Apparent Terminal Elimination Rate Constant (Lambda [z]) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Apparent Initial Half-life (t[1/2alpha]) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The t(1/2alpha) is defined as 0.693/Lambda (alpha).
Apparent Terminal Half-life (t[1/2term]) of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 | Pre-dose; 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
  The t(1/2term) is defined as 0.693/Lambda (z).
Amount of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 excreted in Urine (Ae[x-y]) | Up to 48 hours post-dose
  Amount excreted into urine over a given time interval, calculated from the urinary drug concentration of the collection interval x to y hours post dosing multiplied with the associated urine volume of the interval.
Total Amount of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 excreted in Urine (Ae[total]) | Up to 48 hours post-dose
  Total amount excreted into urine, calculated by adding the amounts of the individual intervals together {Ae[0-48hours(h)]}.
Total Percentage of ALS 008176, ALS-008206, ALS-008112, and ALS-008144 dose excreted into urine | Up to 48 hours post-dose
  Total percentage of the dose excreted into urine, calculated as 100 * (Ae[total]/Dose).
Renal clearance | Up to 48 hours post-dose
  Renal clearance calculated as Ae (0-48h)/AUC (0-48h).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (14 days after dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan